CLINICAL TRIAL: NCT00286091
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Phase 3 Study of Denosumab on Prolonging Bone Metastasis-Free Survival in Men With Hormone Refractory Prostate Cancer
Brief Title: Study on Prolonging Bone Metastasis-Free Survival in Men With Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20050147
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: Hormone refractory prostate cancer; androgen independent; ADT; bone metastasis
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injections every 4 weeks during the double-blind treatment phase. Participants then received open-label denosumab 120 mg by subcutaneous injection every 4 weeks during the open-label extension phase.
  Interventions: Biological: Placebo
- Denosumb (Experimental): Participants received 120 mg denosumab administered by subcutaneous injection every 4 weeks during the double-blind treatment phase. Participants then received open-label denosumab 120 mg by subcutaneous injection every 4 weeks during the open-label extension phase.
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: Denosumab — Administered by subcutaneous injection
  Other Names: XGEVA®
  Arms: Denosumb
Biological: Placebo — Same volume subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the treatment effect of denosumab with placebo on prolonging bone metastasis-free survival in men with hormone refractory (androgen independent) prostate cancer who have no bone metastasis at baseline.

DETAILED DESCRIPTION:
Participants were randomized to receive denosumab 120 mg or placebo every 4 weeks (Q4W) until approximately 660 participants developed bone metastasis or died and the primary efficacy and safety analyses were completed.

All participants undergoing scheduled assessments were offered open-label denosumab 120 mg subcutaneous (SC) until they either developed a bone metastasis, obtained access to commercially available product in this setting, or for up to 3 years, whichever came first. For participants who ended participation before the open-label extension (OLE) phase or withdrew from investigational product during the OLE phase, their survival data was to be collected every 6 months for up to 3 years after their last dose of investigational product.

Participants in the Czech Republic and United Kingdom were enrolled under a separate protocol for the OLE phase per Health Authority request, and are reported separately (Study 20080585; NCT01824342).

ELIGIBILITY:
Inclusion Criteria:

* men with histologically confirmed prostate cancer
* bilateral orchiectomy at least 6 months before randomization or continuous androgen-deprivation therapy (ADT) with a gonadotropin releasing hormone (GnRH) agonist or antagonist for at least 6 months before randomization
* total testosterone level less than 50 ng/dL,
* hormone refractory (androgen independent) prostate cancer demonstrated during continuous ADT/post-orchiectomy defined as: 3 consecutive prostate-specific antigen (PSA) values with PSA1 < PSA2 < PSA3, each PSA value must be separated by at least 2 weeks, PSA2 and PSA3 greater than or equal to 1.0 ng/mL,
* high risk for development of bone metastasis defined as PSA value greater than or equal to 8.0 ng/mL, obtained no more than 3 months before randomization OR PSA doubling time less than or equal to 10.0 months

Exclusion Criteria:

* prior or current evidence of radiographically detectable bone metastasis
* known prior or current evidence of any metastatic involvement of distant organs (lymph node metastases in any region is acceptable)
* prior or current intravenous bisphosphonate administration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1435 (Actual)
Dates: Start 2006-01-24 (Actual); Primary Completion 2010-07-30 (Actual); Study Completion 2014-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Smith MR, Saad F, Coleman R, Shore N, Fizazi K, Tombal B, Miller K, Sieber P, Karsh L, Damiao R, Tammela TL, Egerdie B, Van Poppel H, Chin J, Morote J, Gomez-Veiga F, Borkowski T, Ye Z, Kupic A, Dansey R, Goessl C. Denosumab and bone-metastasis-free survival in men with castration-resistant prostate cancer: results of a phase 3, randomised, placebo-controlled trial. Lancet. 2012 Jan 7;379(9810):39-46. doi: 10.1016/S0140-6736(11)61226-9. Epub 2011 Nov 15. PMID 22093187
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects were men ≥ 18 years old with histologically-confirmed, castrate-resistant prostate cancer who were chemically or surgically castrated. The first patient was enrolled into the study on 03 February 2006 and the last patient was enrolled on 23 July 2008.
Pre-assignment Details: Participants were randomized to denosumab or placebo in the double-blind treatment phase. All participants undergoing scheduled assessments were offered open-label denosumab for up to 3 years in the open-label extension phase. Three enrolled patients were excluded from all datasets per ethics committee's instructions due to eligibility violations.
Groups:
- Placebo: Participants received placebo subcutaneous injection every 4 weeks (Q4W) in the double-blind treatment phase. Participants then received open-label denosumab 120 mg by subcutaneous injecton once every 4 weeks for up to 3 years in the open-label extension phase.
- Denosumab: Participants received 120 mg densumab administered by subcutaneous injection every 4 weeks in the double-blind treatment phase. Participants then received open-label denosumab 120 mg by subcutaneous injecton once every 4 weeks for up to 3 years in the open-label extension phase.
Period: Double-blind Treatment Phase
Arm/Group | Placebo | Denosumab
Started | 716 | 716
Received Treatment | 709 (4 participants received ≥ 1 dose of denosumab in error) | 716
On Study at Primary Data Analysis Cutoff | 164 (Primary analysis cut-off date was 30 July 2010) | 174 (Primary analysis cut-off date was 30 July 2010)
Completed | 132 (On study through blinded treatment cutoff date of 09 January 2011) | 123 (On study through blinded treatment cutoff date of 09 January 2011)
Not Completed | 584 | 593
Not completed — Withdrawal by Subject | 103 | 113
Not completed — Protocol-Specified Criteria | 307 | 269
Not completed — Death | 58 | 65
Not completed — Adverse Event | 28 | 40
Not completed — Disease Progression | 22 | 35
Not completed — Other | 25 | 33
Not completed — Administrative Decision | 20 | 21
Not completed — Noncompliance | 8 | 8
Not completed — Lost to Follow-up | 11 | 4
Not completed — Protocol Deviation | 1 | 3
Not completed — Ineligibility Determined | 1 | 2
Period: Open-label Treatment Phase
Arm/Group | Placebo | Denosumab
Started | 110 (Participants in the Czech Republic and UK are reported separately (Study 20080585; NCT01824342)) | 104 (Participants in the Czech Republic and UK are reported separately (Study 20080585; NCT01824342))
Received Treatment | 109 | 101
Completed | 33 (Completed 3 years of open-label treatment) | 33 (Completed 3 years of open-label treatment)
Not Completed | 77 | 71
Not completed — Physician Decision | 24 | 21
Not completed — Adverse Event | 5 | 16
Not completed — Other | 11 | 11
Not completed — Withdrawal by Subject | 14 | 10
Not completed — Death | 10 | 7
Not completed — Disease Progression | 9 | 3
Not completed — Noncompliance | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol-specified Criteria | 1 | 0
Not completed — Missing End of Study Information | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Denosumab | Total
Number analyzed (Participants) | 716 | 716 | 1432
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (8.3) | 73.2 (8.8) | 73.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 716 | 716 | 1432
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 604 | 606 | 1210
  Black or African American | 35 | 41 | 76
  Hispanic or Latino | 37 | 32 | 69
  Asian | 18 | 17 | 35
  Japanese | 2 | 0 | 2
  American Indian or Alaska Native | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 17 | 18 | 35
  Unknown | 0 | 2 | 2
Eastern Cooperative Oncology Group (ECOG)Pperformance Status [Number; unit: participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    Grade 0 | 514 | 505 | 1019
    Grade 1 | 199 | 210 | 409
    Grade 2 | 3 | 1 | 4
    Grade 3 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0
Prostate-Specific Antigen (PSA) Doubling Time [Number; unit: participants]
  ≤ 10 months | 580 | 574 | 1154
  > 10 months | 136 | 142 | 278
Prostate-Specific Antigen (PSA) ≥ 8.0 ng/mL [Number; unit: participants]
  Yes | 471 | 473 | 944
  No | 245 | 243 | 488
Prior Chemotherapy Regimens [Number; unit: participants]
  Yes | 54 | 63 | 117
  No | 662 | 653 | 1315

OUTCOME MEASURES:

1. Primary Outcome: Bone Metastasis-free Survival
Description: The time to the first occurrence of bone metastasis (either symptomatic or asymptomatic) or death from any cause. Participants who did not experience bone metastasis or on-study death were censored at the last on-study contact date or the primary analysis data cutoff date, whichever came first. Median bone metastasis-free survival time was estimated using the Kaplan-Meier method.
Time Frame: From the first dose of investigational product to the primary data cutoff date of 30 July 2010; median time on study was approximately 20 months.
Population: Full analysis set (all randomized participants)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 716 | 716
days | 768.0 [675.00 to 897.00] | 897.00 [773.00 to 1014.00]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Primary and secondary endpoint analyses were conducted hierarchically. To preserve an overall type I error rate of 0.05, a 0.0488 2-sided test of bone metastasis-free survival was performed. If superiority of denosumab over placebo was established, time to first bone metastasis was tested with a 2-sided significance level of 0.050. If superiority of denosumab over placebo was also established, overall survival time was tested at a 2-sided significance level of 0.050; Test type: Superiority or Other; p = 0.0284, Wald test; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.73 to 0.98] — Based on the Cox proportional hazards model stratified by PSA ≥ 8.0 ng/mL, PSA doubling time ≤ 10 months and previous or current chemotherapy for prostate cancer. A hazard ratio < 1 favors denosumab

2. Secondary Outcome: Time to First Bone Metastasis
Description: Time from randomization to the date of first occurrence of bone metastasis (either symptomatic or asymptomatic), excluding death. Participants who did not develop bone metastasis were censored at their last on-study bone assessment date or the primary analysis data cut-off date, whichever was first. Median time to first bone metastasis was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 716 | 716
days | 897.0 [683.00 to 1009.00] | 1010.0 [897.00 to 1156.00]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority or Other; p = 0.0317, Wald test; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.71 to 0.98] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Survival
Description: Time from randomization to the date of death. Participants who were still alive or lost to follow-up by the primary analysis data cut-off date were censored at their last contact date (on-study or during survival follow-up) or the primary analysis data cut-off date, whichever was first.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 716 | 716
days | 1365.0 [1220.00 to NA] — Could not be estimated due to the low number of events at the time of data cut-off | 1335.0 [1221.00 to NA] — Could not be estimated due to the low number of events at the time of data cut-off
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority or Other; p = 0.9125, Wald test; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.85 to 1.20] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Median investigational product exposure was 18.4 and 19.3 months in the placebo and denosumab groups respectively during the double blind phase and 23.7 and 24.9 months during the open-label treatment phase.
Description: Four participants who were randomized to placebo received ≥ 1 dose of denosumab; therefore, these participants were included within the denosumab group for the safety analyses.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- DB: Placebo: Participants received placebo subcutaneous injection every 4 weeks (Q4W) in the double-blind (DB) treatment phase.
- DB: Denosumab 120 mg Q4W: Participants received 120 mg densumab administered by subcutaneous injection every 4 weeks in the double-blind treatment phase.
- OLE: Placebo/ Denosumab 120 mg Q4W: Participants who received placebo in the double-blind treatment phase received open-label denosumab 120 mg by subcutaneous injecton once every 4 weeks for up to 3 years in the open-label extension (OLE) phase.
- OLE: Denosumab/ Denosumab 120 mg Q4W: Participants who received denosumab in the double-blind treatment phase received open-label denosumab 120 mg by subcutaneous injecton once every 4 weeks for up to 3 years in the open-label extension phase.
Arm/Group | DB: Placebo | DB: Denosumab 120 mg Q4W | OLE: Placebo/ Denosumab 120 mg Q4W | OLE: Denosumab/ Denosumab 120 mg Q4W
Serious Adverse Events (participants affected / at risk) | 332/705 | 341/720 | 39/109 | 36/101
Other Adverse Events (participants affected / at risk) | 585/705 | 599/720 | 80/109 | 74/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=705) | DB: Denosumab 120 mg Q4W (N=720) | OLE: Placebo/ Denosumab 120 mg Q4W (N=109) | OLE: Denosumab/ Denosumab 120 mg Q4W (N=101)
Anaemia (Blood and lymphatic system disorders) | 12 | 25 | 2 | 3
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 4 | 0 | 0
Angina pectoris (Cardiac disorders) | 3 | 5 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 4 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 12 | 6 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 2 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 3 | 2 | 1 | 1
Cardiac failure (Cardiac disorders) | 3 | 3 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 7 | 6 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 3 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 2 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 3 | 0 | 0 | 0
Coronary artery thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 2 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 10 | 12 | 4 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 6 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 2 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Trifascicular block (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Syringomyelia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 3 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 3 | 2 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 5 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 4 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Oesophageal rupture (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral mucosa erosion (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 6 | 0 | 0
Rectal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Asthenia (General disorders) | 10 | 9 | 0 | 0
Chest pain (General disorders) | 3 | 4 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 1
Death (General disorders) | 4 | 4 | 1 | 1
Device battery issue (General disorders) | 1 | 0 | 0 | 0
Device malfunction (General disorders) | 1 | 0 | 0 | 0
Device occlusion (General disorders) | 1 | 3 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 1 | 0
General physical health deterioration (General disorders) | 3 | 5 | 0 | 1
Generalised oedema (General disorders) | 1 | 1 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0 | 0
Local swelling (General disorders) | 1 | 1 | 0 | 0
Malaise (General disorders) | 0 | 6 | 0 | 0
Multi-organ failure (General disorders) | 2 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 2 | 0 | 1
Oedema peripheral (General disorders) | 1 | 2 | 1 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 10 | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1 | 0 | 0
Abscess (Infections and infestations) | 1 | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 0 | 0 | 1 | 0
Abscess of salivary gland (Infections and infestations) | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Anal infection (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 2 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 3 | 1 | 0
Cardiac infection (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 4 | 6 | 1 | 2
Chest wall abscess (Infections and infestations) | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium colitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 1 | 0 | 0
Dental fistula (Infections and infestations) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 2 | 1 | 2
Empyema (Infections and infestations) | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Epiglottitis (Infections and infestations) | 1 | 0 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Gingival abscess (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 0
Human ehrlichiosis (Infections and infestations) | 1 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 2 | 0 | 0
Neutropenic infection (Infections and infestations) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 4 | 1 | 0
Osteomyelitis acute (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 1 | 0 | 0
Penile infection (Infections and infestations) | 0 | 1 | 0 | 0
Perineal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Perineal infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 16 | 13 | 2 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 2 | 2 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Scrotal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 8 | 6 | 0 | 1
Septic shock (Infections and infestations) | 1 | 1 | 2 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 15 | 15 | 2 | 3
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 4 | 3 | 0 | 2
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 6 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 8 | 1 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Retinal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspiration bronchial (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0
Laboratory test abnormal (Investigations) | 0 | 1 | 0 | 0
Ultrasound liver abnormal (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 9 | 7 | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 9 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 7 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 12 | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 7 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 10 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0
Metastases to larynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to small intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 15 | 1 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 0 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 10 | 8 | 2 | 2
Cerebrovascular disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Coma (Nervous system disorders) | 0 | 1 | 0 | 0
Complex partial seizures (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 4 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 1
Epilepsy (Nervous system disorders) | 3 | 0 | 0 | 0
Gait apraxia (Nervous system disorders) | 1 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 4 | 8 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 2 | 1 | 1
Vertebral artery occlusion (Nervous system disorders) | 0 | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 4 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 2 | 0 | 0
Anuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 5 | 0 | 0
Bladder dilatation (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 3 | 0 | 0
Bladder neck sclerosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 2 | 1 | 0 | 0
Bladder perforation (Renal and urinary disorders) | 0 | 2 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 3 | 3 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 3 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 3 | 7 | 0 | 0
Haematinuria (Renal and urinary disorders) | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 25 | 37 | 2 | 5
Haemorrhage urinary tract (Renal and urinary disorders) | 2 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 11 | 15 | 0 | 1
Hydroureter (Renal and urinary disorders) | 0 | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 2 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 2 | 2 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 6 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 9 | 16 | 1 | 2
Renal failure acute (Renal and urinary disorders) | 16 | 12 | 4 | 2
Renal failure chronic (Renal and urinary disorders) | 3 | 2 | 1 | 0
Ureteric dilatation (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 4 | 3 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 3 | 2 | 0 | 0
Urethral pain (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 4 | 3 | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 2 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 33 | 56 | 6 | 5
Urinary tract disorder (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 12 | 5 | 1 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 2 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 1 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 3 | 1 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 2 | 0 | 4 | 0
Prostatic perforation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Testicular atrophy (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 0 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 1 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Physical disability (Social circumstances) | 1 | 0 | 0 | 0
Bladder catheterisation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Cancer surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0
Cardioversion (Surgical and medical procedures) | 1 | 0 | 0 | 0
Cataract operation (Surgical and medical procedures) | 2 | 1 | 0 | 0
Colostomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Cystostomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Debridement (Surgical and medical procedures) | 1 | 0 | 0 | 0
Finger amputation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Heart valve operation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0
Orchidectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Skin graft (Surgical and medical procedures) | 1 | 0 | 0 | 0
Stent placement (Surgical and medical procedures) | 1 | 0 | 0 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 2 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Aortic dilatation (Vascular disorders) | 0 | 1 | 0 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 6 | 8 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 3 | 0 | 0
Hypertension (Vascular disorders) | 3 | 3 | 0 | 3
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 4 | 5 | 0 | 1
Intermittent claudication (Vascular disorders) | 1 | 3 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 2 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 1 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 2 | 0 | 0
Thrombosis (Vascular disorders) | 3 | 1 | 1 | 0
Vascular occlusion (Vascular disorders) | 1 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 2 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=705) | DB: Denosumab 120 mg Q4W (N=720) | OLE: Placebo/ Denosumab 120 mg Q4W (N=109) | OLE: Denosumab/ Denosumab 120 mg Q4W (N=101)
Anaemia (Blood and lymphatic system disorders) | 74 | 80 | 12 | 10
Abdominal pain (Gastrointestinal disorders) | 47 | 59 | 3 | 7
Constipation (Gastrointestinal disorders) | 124 | 128 | 13 | 15
Dental caries (Gastrointestinal disorders) | 10 | 16 | 3 | 6
Diarrhoea (Gastrointestinal disorders) | 102 | 110 | 8 | 10
Nausea (Gastrointestinal disorders) | 95 | 98 | 4 | 14
Toothache (Gastrointestinal disorders) | 16 | 32 | 1 | 6
Vomiting (Gastrointestinal disorders) | 55 | 59 | 3 | 10
Asthenia (General disorders) | 91 | 92 | 8 | 11
Fatigue (General disorders) | 82 | 98 | 5 | 8
Oedema peripheral (General disorders) | 88 | 94 | 5 | 11
Bronchitis (Infections and infestations) | 32 | 40 | 3 | 3
Influenza (Infections and infestations) | 38 | 49 | 7 | 6
Nasopharyngitis (Infections and infestations) | 72 | 68 | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 23 | 46 | 8 | 8
Urinary tract infection (Infections and infestations) | 96 | 108 | 15 | 14
Fall (Injury, poisoning and procedural complications) | 42 | 36 | 3 | 3
Weight decreased (Investigations) | 42 | 39 | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 61 | 63 | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 116 | 123 | 11 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 159 | 166 | 24 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 28 | 46 | 6 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 59 | 58 | 8 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 24 | 24 | 6 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 17 | 1 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 88 | 101 | 12 | 10
Pain in jaw (Musculoskeletal and connective tissue disorders) | 7 | 25 | 2 | 6
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 58 | 56 | 0 | 1
Dizziness (Nervous system disorders) | 56 | 63 | 7 | 6
Headache (Nervous system disorders) | 54 | 67 | 3 | 5
Insomnia (Psychiatric disorders) | 44 | 46 | 4 | 2
Dysuria (Renal and urinary disorders) | 66 | 73 | 5 | 7
Haematuria (Renal and urinary disorders) | 90 | 87 | 17 | 11
Nocturia (Renal and urinary disorders) | 26 | 39 | 3 | 3
Pollakiuria (Renal and urinary disorders) | 50 | 61 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 30 | 30 | 8 | 4
Urinary retention (Renal and urinary disorders) | 63 | 73 | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 60 | 55 | 6 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 57 | 61 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 32 | 37 | 2 | 3
Hot flush (Vascular disorders) | 32 | 41 | 1 | 1
Hypertension (Vascular disorders) | 49 | 59 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.